CLINICAL TRIAL: NCT01150487
Title: Paired Bone Marrow Aspirations to Assess the Variability of Allo-ELISPOT and Allo-Specificities Assays in Sensitized Renal Allograft Recipients
Brief Title: Paired Marrow Aspirations to Assess Assays in Sensitized Renal Allograft Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Mark Stegall, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-002572; R21AI125719 (NIH)
Record Dates: First submitted 2010-06-23; First posted 2010-06-25 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Transplantation, Kidney; Living Donors; Kidney Transplant Recipients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kidney recipients or kidney donors (Experimental): Patients who have had a Kidney transplant or are undergoing a kidney transplant. Kidney donors.
  Interventions: Procedure: bone marrow aspirations; Procedure: lymph node collection

INTERVENTIONS:
Procedure: bone marrow aspirations — A bone marrow aspiration from each hip bone of the patients.
Procedure: lymph node collection — An Iliac lymph node collection.

SUMMARY:
The aim of this study is to determine a comprehensive immune profile of transplant donors and recipients through assessment of immune cell compositions in bone marrow, and lymph nodes.

DETAILED DESCRIPTION:
The aim of this risk protocol is to determine the variability of the AlloElispot and Allospecificities assay.

Our group has developed a number of assays to assess the immune cell population in our transplant population. This has included: 1) the number of donor-specific alloantibody (DSA) secreting bone marrow derived plasma cells (AlloELISPOT assay), 2) the function of DSA-secreting Plasma cells (Allospecificities assay), 3)Culture of plasma cells in human stromal cells to produce specific HLA antibodies and tetanus antibodies, 4) Understand the critical pathways for the survival and function of plasma cells, 5)Characterize the different phenotypes and genotypes of the plasma cell, 6)Phenotype analyses of the immune cell population using flow cytometry and/or mass spectrometry (ie. cytometry by time of flight/CyTOF), 7)Functional assessments of T and B-cells, and 8)T-cell receptor diversity.

These assays were developed over the years and already have provided an important means of testing new therapeutic protocols aimed at controlling DSA production. It is important to note that repeated attempts to isolate PCs from peripheral blood have been unsuccessful (PCs are extremely rare in peripheral blood) and the bone marrow is the only accessible source of PCs.

It is now clear to that we have reached a point that we must validate these assays (coefficient of variation, etc), in order to appropriately evaluate data derived from these assays. Inter-assay variability can be assessed by performing two paired assays in the same patient. This could be done in two ways-paired bone marrow aspirations separated by time or two bone marrow aspirations performed at the same time. We have decided to pursue the latter approach. We will do both marrows either at the time of transplantation or while they are undergoing a surgical procedure. Lymph node retrieval will also be performed at the time for abstraction of immune cells for additional analysis. We believe that this is safe and will be well-tolerated and will provide the data that we need to validate the assays.

ELIGIBILITY:
Inclusion criteria.

* Pre or post renal transplant recipients.
* Renal transplant donors.
* Those who give voluntary written informed consent before performance of any study-related procedures, which are not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion criteria.

* Any patient currently receiving systemic anticoagulation therapy with heparin or coumadin.
* Patient has a platelet count of <30 x 10(9)/L within 14 days before enrollment.
* Patient has an absolute neutrophil count of ANC<1.0 x 10(9)/L within 14 days before enrollment.
* Patient has received other investigational drugs within14 days before enrollment.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for malignancy within 5 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Contraindication to kidney transplantation or donation-active infection, comorbid medical conditions, etc

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2010-10-05 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
To determine a comprehensive immune profile of transplant donors and recipients through assessment of immune cell compositions in bone marrow, and lymph nodes. | 1 week Post bone marrow and lymph node collection.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stegall, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No